CLINICAL TRIAL: NCT06841809
Title: The Role of Radiographic Indices in the Evaluation of Hand and Wrist Pathologies in Patients With Carpal Tunnel Syndrome
Brief Title: Analysis of Radiographic Indices in Carpal Tunnel Syndrome
Status: Completed | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nadide Koca, Principal Investigator, Ankara Training and Research Hospital
Other Study IDs: AnkaraTRH-FTR-NK-03
Record Dates: First submitted 2025-02-16; First posted 2025-02-24 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-05

CONDITIONS: Carpal Tunnel Syndrome (CTS); Wrist; X-Ray; Radiography
Keywords: Carpal Tunnel Syndrome (CTS); wrist; X-Ray
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case: Patients referred to the EMG clinic and diagnosed with carpal tunnel syndrome were selected. All of these patients underwent bilateral EMG.
- Control: The control group was randomly selected from patients who applied with other hand and wrist complaints during the same period and who had wrist radiographs, and who were matched with the study group in terms of age and gender.

SUMMARY:
The aim of this study was to compare wrist radiographic indices in patients with idiopathic carpal tunnel syndrome (CTS) with normal cases. The investigators believe that the investigators can contribute to the development of new treatment strategies by determining the radiographic features that contribute to the development of CTS.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common mononeuropathy of the upper extremity. It occurs as a result of compression of the median nerve in the carpal tunnel during its course in the wrist. Clinical symptoms are characterized by numbness and tingling in the first 3 fingers and the radial half of the 4th finger, which are compatible with the distribution of the median nerve. Electrophysiologically, it is classified as mild, moderate and severe. As the disease duration increases, atrophy and weakness may develop in the thenar muscles. The incidence is 4-5% worldwide and is more common in women between the ages of 40-60.

Pathophysiology consists of mechanical compression, increased pressure, ischemia in the median nerve and local metabolic changes.

Among the risk factors, occupations that require repeated flexion and extension of the wrist constitute environmental risk factors. Extension can increase the tunnel pressure by 10 times, while flexion can increase it by more than 8 times. Systemic risk factors for CTS are pregnancy, menopause, obesity, renal failure, hypothyroidism, oral contraceptive use, and congestive heart failure.

Diabetes, alcoholism, vitamin deficiency or toxicity, and exposure to toxins are neuropathic risk factors. Localized risk factors include mass lesions that compress the tunnel, arthritis, and radius distal end fractures.

Despite these risk factors, most cases of CTS are still classified as idiopathic.

CTS often develops in the late period after radius distal end fractures. The mechanism here is multifactorial and includes malunion, chronically inflamed synovium, volar callus, and scar tissue. However, in late CTS cases developing after Colles fractures, it has been determined that carpal alignment is greatly affected by the displacement of the radius.

This finding has drawn the attention of researchers to the radiographic features of the distal radius and carpal bone in the etiopathogenesis of idiopathic CTS.

There are several studies conducted on wrist radiographic features in idiopathic CTS.

In a case-control study evaluating the radiographic parameters of 94 wrists of 62 idiopathic carpal tunnel syndrome patients and 94 asymptomatic wrists of 94 controls, radial inclination, volar inclination, ulnar variance and transverse and anteroposterior diameters were measured on posteroanterior and lateral radiographs of the wrist. The measurements were made by two evaluators and the average of the measurements of the two was taken. At the end of this study, a significant difference was found only in ulnar variance and it was reported that positive ulnar variance may be an index to be considered in CTS.

In another study, wrist radiographs of 75 idiopathic CTS patients who underwent carpal tunnel release surgery were compared with the radiographs of 87 normal control group participants. Radial inclination, volar inclination, ulnar variance, radiolunate angle (RLA) and lunate-radius axis distance were measured. Data were measured using two independent raters and the average of these measurements was taken. RLA and lunate-radius axis distance were found to be significant between the two groups. The researchers concluded that excessive dorsiflexion and volar displacement of the lunate can be considered as CTS risk factors.

In another study conducted on female patients with CTS, radiographs of 55 CTS hands of 40 female patients were compared with healthy control subjects. Capitate length, Carpal height, Palm length, Scaphoid-Pisiform Width Index (SPWI) and Palmar ratio values were found to be lower in the patient group. The researchers reported that the carpal bone configuration affects the proximal part of the carpal tunnel and may affect the compression of the median nerve in female patients.

The purpose of this study; to compare the radiographic features of the wrist of patients with idiopathic CTS with the radiographic features of normal control cases. For this purpose, the investigators examined the radiographic features of the distal radius and the scaphoid and lunate bones, which are the two bones that articulate with it and also participate in the posterior proximal floor of the carpal tunnel. The investigators also evaluated whether radiographic features are related to the severity of CTS and symptom severity. The investigators believe that the results to be obtained will contribute to treatment strategies. This study is the first to investigate the relationship between the radioscaphoid angle (RSA), scapholunate angle (SLA) and radiographic indices and symptoms in idiopathic carpal tunnel syndrome (CTS).

ELIGIBILITY:
Inclusion Criteria:

* Not having had any previous surgical procedures on the hand or wrist
* Not having had a major hand or wrist trauma
* No structural disorders in the bone structure

Exclusion Criteria:

* Being under 18 years of age
* History of major hand-wrist trauma or surgery
* Acromegaly
* Rheumatoid arthritis
* Systemic lupus erythematosus
* GUT arthritis
* Psoriatic arthritis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The case group will consist of patients referred to the EMG clinic and diagnosed with carpal tunnel syndrome (CTS). All of these patients will undergo bilateral EMG. The control group was randomly selected from patients with hand and wrist complaints, who were matched with the study group in terms of age and gender, and who had hand complaints other than CTS.
Sampling Method: Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2025-02-16 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Measurement of Radiographic Indices | up to 12 weeks
  Radio-lunate Angle (RLA): The distance between the tangential line connecting the two distal poles of the lunate root and the line drawn perpendicular to the central medullary canal of the distal radius.

SECONDARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire | up to 12 weeks
  The Boston Carpal Tunnel Syndrome Questionnaire (BCTSQ) is specifically designed for people with carpal tunnel syndrome (CTS) and provides insight into symptoms and severity when performing specific actions. Normal 24-hour periods are measured over the past 2 weeks.
  The BCTSQ consists of two separate scales: the Symptom Severity Scale (SSS), which consists of 11 questions, and the Functional Status Scale (FSS), which consists of 8 items and requires participants to rate the difficulty of each item on a five-point scale. A final score is calculated for each scale (the sum of individual scores divided by the number of items) and ranges from 1 to 5, with a higher score indicating more severe disability.
Electromyography Examination | up to 12 weeks
  Electromyography (EMG), which is electromyography, is a diagnostic method used to determine the health status of muscles and motor neurons that control muscles.
  Upper extremity nerve conduction studies were performed using supramaximal percutaneous stimulation with a constant current stimulator and surface electrode recording.
  Mild CTS: The difference between the median sensory response distal latency and the ulnar sensory response distal latency is > 1 msec or the difference between the median-ulnar nerve peak latencies recorded at the 4th finger is > 0.5 msec Moderate CTS: In addition to the above, the distal latency of the median motor nerve is prolonged (> 4.0 msec) Severe CTS: Frequently low/absent sensory potential amplitude and decreased motor response amplitude (< 5.0 mV) or delayed latency (> 5.5 msec).
Measurement of Radiographic Indices | up to 12 weeks
  Radial Inclination (RE): The angle between a line connecting the radial styloid tip and the ulnar aspect of the distal radius and a second line perpendicular to the longitudinal axis of the radius.
Measurement of Radiographic Indices | up to 12 weeks
  Volar Inclination (VE): The angle of the distal radial surface relative to the vertical shaft line. It is evaluated on the lateral radiograph.
Measurement of Radiographic Indices | up to 12 weeks
  Carpal Height Ratio (CHR): It is found by measuring the height of the carpal bones vertically and dividing it by the length of the 3rd metacarpal.
Measurement of Radiographic Indices | up to 12 weeks
  Wrist Anteroposterior Diameter (APD): The distance between the volar and dorsal edges of the distal radius.
Measurement of Radiographic Indices | up to 12 weeks
  Transfers Diameter (TC): The distance between the radial edge of the radius and the ulnar edge of the ulna at the level of the radiocarpal joint.
Measurement of Radiographic Indices | up to 12 weeks
  Ulnar Variance (UV): The vertical distance between the articular surface of the ulna head and the lunate facet of the distal radius.
Measurement of Radiographic Indices | up to 12 weeks
  Radio-scaphoid Angle (RSA): The angle between the tangential line connecting the palmar proximal and distal edges of the scaphoid and the line drawn to the central medullary canal of the distal radius.
Measurement of Radiographic Indices | up to 12 weeks
  Scapholunate Angle (SLA): The angle between the longitudinal axes of the lunate and scaphoid on a lateral radiograph.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Training and Research Hospital, University of Health Sciences, Department of Physical Therapy and Rehabilitation, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uysal T, Ramoglu SI, Basciftci FA, Sari Z. Chronologic age and skeletal maturation of the cervical vertebrae and hand-wrist: is there a relationship? Am J Orthod Dentofacial Orthop. 2006 Nov;130(5):622-8. doi: 10.1016/j.ajodo.2005.01.031. PMID 17110259
- [Background] Ferreira Branco D, Bouvet C, Hamard M, Beaulieu JY, Poletti PA, Boudabbous S. Reliability of radio-ulnar and carpal alignment measurements in the wrist between radiographs and 3D imaging. Eur J Radiol. 2022 Sep;154:110417. doi: 10.1016/j.ejrad.2022.110417. Epub 2022 Jun 22. PMID 35772337
- [Background] Garcia-Elias M, An KN, Amadio PC, Cooney WP, Linscheid RL. Reliability of carpal angle determinations. J Hand Surg Am. 1989 Nov;14(6):1017-21. doi: 10.1016/s0363-5023(89)80053-x. PMID 2584642
- [Background] Okan N, Caboglu F, Mertoglu T, Durakbasa O, Gorgec M. [The measurement of wrist kinematics in children 4 to 16 years old and the comparison of the scapholunate distance with adult values]. Acta Orthop Traumatol Turc. 2004;38(1):30-3. Turkish. PMID 15054295
- [Background] Wang YC, Tseng YC, Chang HY, Wang YJ, Chen CJ, Wu DY. Gender differences in carpal height ratio in a taiwanese population. J Hand Surg Am. 2010 Feb;35(2):252-5. doi: 10.1016/j.jhsa.2009.11.010. PMID 20141895
- [Background] Vaezi T, Hassankhani GG, Ebrahimzadeh MH, Moradi A. Evaluation of Normal Ranges of Wrist Radiologic Indexes in Mashhad Population. Arch Bone Jt Surg. 2017 Nov;5(6):451-458. PMID 29299502
- [Background] Ar Altamimi A, Gharaibeh MA, Shokor MA, Dawod MS, Alswerki MN, Al-Odat OM, Elkhaldi RH. Association between carpal height ratio and ulnar variance in normal wrist radiography. BMC Musculoskelet Disord. 2024 Jul 9;25(1):524. doi: 10.1186/s12891-024-07647-z. PMID 38982384
- [Background] Taillac H, Holzgrefe R, Hao KA, Hones KM, Wright TW, King JJ, Satteson E, Matthias RC. Intercarpal Angles on Hand Versus Wrist Films: Are Hand Radiographs Sufficient for Assessing Intercarpal Angles? J Hand Surg Am. 2024 Dec;49(12):1273.e1-1273.e6. doi: 10.1016/j.jhsa.2023.04.012. Epub 2023 May 27. PMID 37245153
- [Background] Sarhan MY, Altamimi AA, Gharaibeh MA, Akel A, Abu Shokor M, Salem OA, Balbisi B, Abu-Jeyyab M. Evaluation of Normal Ranges of Wrist Radiologic Indexes in Jordanian Population. Orthop Rev (Pavia). 2024 Aug 3;16:120049. doi: 10.52965/001c.120049. eCollection 2024. PMID 39105053
- [Derived] Koca N, Nazligul NK. Evaluation of wrist radiographic indices in people with idiopathic carpal tunnel syndrome: a prospective cross-sectional study. Ann Phys Rehabil Med. 2026 Jan 8;69(2):102068. doi: 10.1016/j.rehab.2025.102068. Online ahead of print. PMID 41512671